CLINICAL TRIAL: NCT05488210
Title: Study to Evaluate the Effect of Consuming an Oral Nutritional Supplement (ONS) Specifically for Diabetic Patients on Adherence and Gastrointestinal Tolerance and Nutritional Status in Patients With DM2 and Malnutrition
Brief Title: Study About Adherence and Tolerance of an Oral Nutritional Supplement (ONS) Specific for Diabetic Patient.
Acronym: DIABEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Fundació Eurecat (Other); Laboratoires Grand Fontaine S.L (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI-6092
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-04

CONDITIONS: Diabetes; Malnutrition
Keywords: DM2; Oral nutritional supplement; Malnourished
MeSH Terms: conditions — Diabetes Mellitus; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malnourished DM2 patients: Diabetic patients who present malnutrition through the GLIM criteria
  Interventions: Dietary Supplement: FontActiv DiaBest HP/HC

INTERVENTIONS:
Dietary Supplement: FontActiv DiaBest HP/HC — Daily intake of two FontActiv DiaBest HP/HC during 2 months
  Other Names: Experimental

SUMMARY:
Diabetes Mellitus (DM) is one of the most prevalent chronic diseases today, it is reaching epidemic proportions, mainly caused by the increase in type 2 diabetes (DM2).The foundation of any hypoglycemic treatment is based on a healthy diet, daily physical exercise and adequate health education with the collaboration of the patient. Diet is sometimes the only necessary therapy since approximately 80% of patients with DM2 are usually overweight, what is mainly wanted with diet is to achieve normal blood glucose levels both fasting and in the postprandial phase. This diet must be a varied diet combining foods from the different food groups; however, carbohydrate control must be one of the key strategies for glycemic control. Currently, there is also talk of the concept of disease-related malnutrition (DRM). DRM is malnutrition associated with a pathological state, with the presence of inflammation being a key factor in determining its etiology. This inflammation can be chronic or acute depending on the type of pathology. Therefore, the fiber and carbohydrate composition of oral nutritional supplements are important for glycemic control, so a study is proposed to evaluate the effect of consuming a ONS hypercaloric/high-protein (HC/HP) with fiber, and enriched in calcium, Vitamin D and DHA on adherence and tolerance of the product and nutritional status in patients with DM2 and malnutrition.

DETAILED DESCRIPTION:
Longitudinal, prospective exploratory study, to evaluate the effect of consuming an oral nutritional supplement (ONS) HC/HP with fiber, and enriched in calcium, Vitamin D and Docosahexaenoic acid (DHA) on adherence and tolerance of the product and nutritional status in patients with DM2 and malnutrition, in a period of 60 days. Twenty-four volunteers will be recruited at the La Paz University Hospital of Madrid. Participants should meet the next inclusion criteria: men and woman enter 18 and 85, with DM2 previously diagnosed and controlled, with malnutrition diagnosed according to the Global Leadership Initiative on Malnutrition (GLIM) criteria, who require taking ONS, willing to consume the ONS during the study and adequate cultural level and understanding of the clinical study. Follow up will include 4 individualized visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women enter 18 and 85 years old.
* Patients with DM2 previously diagnosed and controlled.
* Patients with malnutrition diagnosed according to GLIM criteria.
* Patients who require taking ONS.
* Patients willing to consume the ONS during the study period.
* Patients with adequate cultural level and understanding of the clinical study.
* Patients who agree to voluntarily participate in the study and who give their informed consent in writing.

Exclusion Criteria:

* Subjects with enteral or parenteral nutrition.
* Subjects with poorly controlled DM2.
* Subjects with dementia, eating behavior disorders, history of serious neurological or psychiatric pathology that may interfere with adherence to the consumption of the ONS.
* Subjects suffering from alcoholism or substance abuse that may interfere with adherence to the consumption of the ONS.
* Subjects with a diagnosis of kidney or liver disease under pharmacological treatment.
* Subjects with infections or any condition that interferes with nutrient digestion, absorption, metabolism, or excretion (including gastroparesis).
* Subjects with chronic gastrointestinal diseases that affect the digestion or absorption of nutrients.
* Subjects with allergies or intolerances to any of the ingredients of the formula.
* Subjects with socio-family problems that prevent them from participating in the study.
* Pregnant or lactating women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients who present malnutrition through the GLIM criteria
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Weight gain (kg) | Day 0, Day 60
  Changes in body weight. It is measured using a digital scale for clinical use (capacity 0-150 kg),with the person positioned with their back to the viewer, without shoes, wearing a minimum of warm clothing (pants and t-shirt), heels together, looking forward and posture straight body.
Fat mass (%) | Day 0, Day 60
  Changes in the percentage (%) of Fat Mass via bioelectrical impedance
Muscle mass (%) | Day 0, Day 60
  Changes in the percentage (%) of Muscle Mass via bioelectrical impedance

SECONDARY OUTCOMES:
Waist circumference (cm) | Day 0, Day 60
  The subject assumes a position with arms crossed at the chest. The perimeter is taken at the narrowest level, between the lower costal margin (10th rib) and the iliac crest. The anthropometrist stands in front of the subject, who has his arms slightly abducted, to allow the waist to run around the abdomen. Values greater than 80 centimeters (women) and 94 centimeters (men) are considered a risk for cardiovascular diseases.
Body Mass Index (kg/m2) | Day 0, Day 60
  It is the relationship between the individual's body weight (kg) and height (m) squared: Weight/Height2. Values greater than 24,9 kg/m2 are considered as overweight
Extracellular water (%) | Day 0, Day 60
  Changes in the percentage (%) of Extracellular Water via bioelectrical impedance
Intracellular water (%) | Day 0, Day 60
  Changes in the percentage (%) of Intracellular Water via bioelectrical impedance
Total Body Water (%) | Day 0, Day 60
  Changes in the percentage (%) of Total Body Water via bioelectrical impedance
Phase angle (º) | Day 0, Day 60
  Changes in the phase angle (grades) via bioelectrical impedance
Body Cell Mass (%) | Day 0, Day 60
  Changes in the percentage (%) of Body Cell Mass via bioelectrical impedance
Albumin serum concentration (g/dL) | Day 0, Day 60
  Changes in serum albumin concentration. The normal range is 3.4 to 5.4 g/dL (34 to 54 g/L)
Prealbumin serum concentration (mg/dL) | Day 0, Day 60
  Changes in serum prealbumin concentration. Normal results in adults range between 15 and 36 milligrams per deciliter (mg/dL) or 150 and 360 milligrams per liter (mg/L)
Glucose serum concentration (mg/dL) | Day 0, Day 60
  Changes in fasting serum glucose concentration. The levels are between 74 and 100 mg/dL.
Insulin serum concentration (IU/mL) | Day 0, Day 60
  Changes in serum insulin levels. A basal insulin level between 5-25 IU/ml is considered normal, higher than 30 U/ml suggests insulin resistance. Insulin maximum value 6 to 8 times the basal value.
HbA1c serum concentration (%) | Day 0, Day 60
  Changes in the percentage of HbA1c. An HBA1c level of less than 5.7% is normal, 5.7 to 6.4% indicates prediabetes, and 6.5 or greater indicates diabetes. Within the prediabetes range (5.7 to 6.4%), the higher the A1c value, the greater the risk of developing type 2 diabetes
Total Cholesterol serum concentration (mg/dL) | Day 0, Day 60
  Changes in total cholesterol concentration. A concentration less than 200 mg/dL is recommended, with a normal upper limit between 200 and 239 mg/dL. Measurements above 240 mg/dL indicate excessive consumption through diet or familial hypercholesterolemia
Triglycerides serum concentration (mg/dL) | Day 0, Day 60
  Changes in triglyceride concentration. Normal values are less than 150 mg/dL; the upper limit is between 150 and 199 mg/dL. However, values between 200 and 499 mg/dl are considered high or very high (above 500 mg/dl).
LDL-cholesterol serum concentration (mg/dL) | Day 0, Day 60
  Changes in LDL-cholesterol concentration. Optimal levels are less than 100 mg/dL, although concentrations between 100 and 129 mg/dL are considered almost optimal. The upper limit of normal is between 130 and 159. Values between 160 and 189 mg/dL are considered high, and those above 190 mg/dL as very high.
HDL-cholesterol serum concentration (mg/dL) | Day 0, Day 60
  Changes in HDL-cholesterol concentration. Values above 60 mg/d Lare considered a protective factor against cardiovascular diseases.Concentrations between 40 and 59 mg/dL are correct, while values below 40 mg/dL are one of the main risk factors for cardiovascular disease.
Creatinine serum concentration (mg/dL) | Day 0, Day 60
  Changes in creatinine concentration. Normal values are 0.7 to 1.3 mg/dL (61.9 to 114.9 µmol/L) for men and 0.6 to 1.1 mg/dL (53 to 97.2 µmol/L) for women. Women often have lower creatinine levels than men, due to less muscle mass.
Urate serum concentration (mg/dL) | Day 0, Day 60
  Changes in urate concentration. Normal values are between 3.5 and 7.2 milligrams per deciliter (mg/dL).
Adherence to the Mediterranean Diet | Day 0, Day 60
  Questionnaire on Consumption Adherence to the Mediterranean Diet. The questionnaire consists of 14 questions with a variable score on different aspects of the diet and the Mediterranean pattern. A score less than 9 indicates poor adherence, while a score of 9 or more points indicates good adherence.
24 hour food record questionnaire | Day 0, Day 60
  Questionnaire to find out the nutritional and dietary habits of each participant. The volunteer will write down all the food and drinks ingested over 1 day (24 hours). The answers will allow calculating the total amount of food consumed and calories ingested. In addition, the data will be evaluated quantitatively and qualitatively, classifying the diet in terms of diversity and balance following the recommendations of the Spanish Society of Community Nutrition (SENC 2016).
International Physical Activity Questionnaire (IPAQ) | Day 0, Day 60
  The questionnaire is divided into 4 categories of questions depending on the type of activity for which information is requested (vigorous, moderate, walking, sedentary). The quantitative results allow calculating the TOTAL Energy Metabolism Rate (MET) x minute/week for each subject. Qualitative results categorize the volunteers' physical activity into low activity (1), moderate activity (2), or vigorous activity (3).
Questionnaire on quality of life (EuroQoL 5D) | Day 0, Day 60
  The EuroQol 5D quality of life questionnaire will be used. The questionnaire is divided into two parts. In the first, questions are asked regarding mobility, personal care, daily activities and the presence of pain, discomfort, anxiety or depression. In the second part, the patient must use a visual analog health scale from 1 to 10 to indicate their subjective state of health, with 0 being the worst state of health imaginable and 10 being the best state of health imaginable.
Gastrointestinal symptoms rating scale (GSRS) | Day 0, Day 60
  The GSRS is a specific instrument for the assessment of digestive symptoms that includes 15 items grouped into 5 blocks based on the different gastrointestinal symptoms. The 5 groups of symptoms represent reflux, abdominal pain, indigestion, diarrhea and constipation. It has a score based on a Likert-type scale of 7 degrees, where 1 represents the most positive option and 7 the most negative.
Sensory perception | Day 0, Day 60
  The taste and olfactory sensory perception of the participants for the products will be evaluated by means of a questionnaire using Visual Analogue Scales (VAS) with a score of 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Samara Palma-Milla, MD, PhD, Principal Investigator — Hospital La Paz
Locations (1):
- Samara Palma Milla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No